CLINICAL TRIAL: NCT02490839
Title: Efficacy of High-dose Dual Therapy Versus Bismuth-containing Quadruple Therapy for Rescue Treatment of Helicobacter Pylori Infection - A Prospective, Randomized, Comparative Study
Brief Title: Efficacy of High-dose Dual Therapy vs Bismuth-containing Quadruple Therapy for Rescue Treatment of Hp Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201504037MINB
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; high dose dual therapy; bismuth-containing quadruple therapy; antibiotic resistance
MeSH Terms: interventions — Rabeprazole; Amoxicillin; Proton Pump Inhibitors; Anti-Bacterial Agents; Metronidazole; Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High-dose dual therapy (Experimental): group A-high-dose dual therapy ( rabeprazole 20 mg, tablet, qid + amoxicillin 750 mg, capsule, qid for 14 days)
  Interventions: Drug: High-dose dual therapy (rabeprazole, amoxicillin)
- Bismuth-containing quadruple therapy (Active Comparator): group B-bismuth-containing quadruple therapy (rabeprazole 20 mg, tablet, bid + tripotassium dicitrate bismuthate 300 mg, tablet, qid + metronidazole 250 mg, tablet, qid + tetracycline 500 mg qid, capsule, for 10 days)
  Interventions: Drug: Bismuth-containing quadruple therapy (rabeprazole, tripotassium dicitrate bismuthate, metronidazole, tetracycline)

INTERVENTIONS:
Drug: High-dose dual therapy (rabeprazole, amoxicillin) — High-dose dual therapy ( rabeprazole 20 mg qid + amoxicillin 750 mg qid for 14 days)
  Other Names: Proton pump inhibitor, Rabeprazole, Pariet®; Antibiotics, Amoxicillin ,Amoxicillin®
  Arms: High-dose dual therapy
Drug: Bismuth-containing quadruple therapy (rabeprazole, tripotassium dicitrate bismuthate, metronidazole, tetracycline) — Bismuth-containing quadruple therapy (rabeprazole 20 mg bid + tripotassium dicitrate bismuthate 300 mg qid + metronidazole 250 mg qid + tetracycline 500 mg qid for 10 days)
  Other Names: Proton pump inhibitor, Rabeprazole, Pariet®; Antibiotics, Metronidazole, Flagyl®; Antibiotics, Tetracycline, Tetracycline®; Colloidal Bismuth, Tripotassium dicitrate bismuthate, KCB®
  Arms: Bismuth-containing quadruple therapy

SUMMARY:
Up to now, there is few randomized, large scale study prospectively and simultaneously comparing the efficacy, adverse effects and patient adherence of high-dose dual therapy (HDDT) and bismuth-containing quadruple therapy (BQT) as rescue regimens for H. pylori eradication.

The aims of this study are:

1. to compare the efficacy of HDDT, and BQT as rescue regimen in H. pylori eradication;
2. to compare the patient adherence and adverse effects of these treatment regimens;
3. to investigate factors that may influence H. pylori eradication by these treatment regimens.

DETAILED DESCRIPTION:
Participants, aged ≥ 20, having H. pylori-positive chronic gastritis with/without peptic ulcers (duodenal or gastric ulcers) will be recruited. All undergo endoscopy with biopsy for rapid urease teat, histology, and bacterial culture before treatment. Four to eight weeks after termination of treatment, H. pylori infection status will be examined by the 13C-urea breath test. The CYP2C19 genotype of each participant will be analyzed by the polymerase chain reaction-based restriction fragment length polymerase (PCR-RFLP) method. A computed generated random numbers sequence will be blocked into two subgroups, say A, and B.

If the patients failed anti-H. pylori therapy previously, they will be invited to enter this study for evaluating the efficacy of these rescue regimens. Participant who meet the inclusion criteria and do not have any one of the exclusion criteria will be randomized to receive one of the following regimens:

group A- HDDT (rabeprazole 20 mg qid + amoxicillin 750 mg qid for 14 days);

group B- BQT ( rabeprazole 20 mg qid + tripotassium dicitrate bismuthate 300 mg qid + metronidazole 250 mg qid + tetracycline 500 mg qid for 10 days);

All participants will be asked to complete a questionnaire and to record symptoms and drug consumption daily during the treatment period. Post-treatment, the participants will be followed up at the Outpatients Clinic to investigate patient adherence and adverse effect of treatment.

ELIGIBILITY:
Inclusion criteria:

1. Participants having H. pylori related chronic gastritis with/without peptic ulcers who are aged greater than 20 years old and are willing to received eradication therapy.

Exclusion criteria:

1. pregnant or nursing woman
2. serious concomitant illness and malignant tumor of any kind
3. history of hypersensitivity to test drugs
4. serious bleeding during the course of the ulcer
5. previous gastric surgery
6. receiving bismuth salts, PPIs, or antibiotics in the previous month.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
The eradication rates as a measure of the efficacy of HDDT, and BQT | 3.5 years
  The eradication rates (efficacy) will be evaluated by intention-to-treat (ITT) and per-protocol (PP) analysis.

SECONDARY OUTCOMES:
Number of participants with adverse effects as a measure of safety | 3.5 years
  The safety will be evaluated by counting the number of participant with adverse events.
Amount of unused medication post treatment as a measure of patient adherence. | 3.5 years
  The patient adherence will be evaluated by counting unused medication after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Chin Yang, M.D.Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan